CLINICAL TRIAL: NCT02053896
Title: A Phase 2 Multi-Center, Open-Label, Switch-Over Trial to Evaluate the Safety and Efficacy of ISU302 in Patients With Type 1 Gaucher Disease Previously Treated With Imiglucerase
Brief Title: A Switch-Over Study of the Safety and Efficacy of ISU302 in Patients With Type 1 Gaucher Disease
Status: Completed | Type: Observational
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISU302-003
Record Dates: First submitted 2014-01-26; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Gaucher Disease
Keywords: Type I Gaucher; ISU302; Imiglucerase
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ISU302: 15~60U/kg (once every 2 weeks for 6 months)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ISU302 in patients with Type 1 Gaucher disease previously treated with Imiglucerase.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with type-1 Gaucher disease
* Patient who was stably treating Gaucher disease with Cerezyme® and who was maintaining the usage and dosage of Cerezyme® for at least 6 months prior to study drug administration
* Patient aged 2 years or higher
* Female patient with contraception during the study period (oral or injectable contraceptive hormones, intrauterine device, physical devices using condom, sponge form, jelly, and femidom, and abstinence)
* Patient who signed the informed consent form after hearing the detailed explanation about this study

  * Definition of the stable treatment of type-1 Gaucher disease:
* No neurologic deficit
* Normal hemoglobin concentration, and platelet count that has increased to ≥100,000/㎣, or maintained to 100,000/㎣
* Normal or no deteriorated bone mineral density
* Normal or no deteriorated splenomegaly or hepatomegaly

Exclusion Criteria:

* Patient who participated in other clinical studies within 90 days before study drug administration
* Patient with unstable hemoglobin and platelet counts for at least 6 months before study drug administration
* Patient with hypersensitivity to Cerezyme®
* Patient positive to HIV antibody, hepatitis B antigen, and hepatitis C antibody
* Patient with Fe, folic acid, or vitamin B12-deficcient anemia
* Patient who received miglustat within 6 months before study drug administration
* Patient who received erythrocyte growth factor or chronic systemic corticosteroids within 6 months before study drug administration
* Patient who had clinically significant splenic obstruction within 12 months before study drug administration
* Pregnant or lactating patient
* Patient who had serious concurrent diseases such as infectious diseases or drug-addicted patient
* Patient who was considered inappropriate for this study by the investigators or sub-investigators

Ages: 8 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient diagnosed with type-1 Gaucher disease
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From Screening to Week 24
  To evaluate the safety of ISU302 in patients with Type 1 Gaucher disease previously treated with Cerezyme® after administering ISU302 alternative to Cerezyme®

SECONDARY OUTCOMES:
Pharmacokinetics | From Screening to Week 24
  Measurement of blood glucocerebrosidase activity for pharmacokinetic assessment after initial study drug administration
hemoglobin concentration | From Screening to Week 24
  Change in hemoglobin concentration
platelet count | From Screening to Week 24
  Change in platelet count
liver and spleen volumes and liver function | From Screening to Week 24
  Changes in liver and spleen volumes and liver function
biomarker levels | From Screening to Week 24
  Changes in biomarker levels (Acid Phosphatase, Angiotensin Converting Enzyme, and Chitotriosidase)
skeletal status and bone mineral density | From Screening to Week 24
  Changes in skeletal status and bone mineral density

REFERENCES:
- [Derived] Choi JH, Lee BH, Ko JM, Sohn YB, Lee JS, Kim GH, Heo SH, Park JY, Kim YM, Kim JH, Yoo HW. A phase 2 multi-center, open-label, switch-over trial to evaluate the safety and efficacy of Abcertin(R) in patients with type 1 Gaucher disease. J Korean Med Sci. 2015 Apr;30(4):378-84. doi: 10.3346/jkms.2015.30.4.378. Epub 2015 Mar 19. PMID 25829804